CLINICAL TRIAL: NCT02774850
Title: Home or Away From Home: Comparing Clinical Outcomes Relevant to the Care of Pediatric Acute Myeloid Leukemia During Periods of Neutropenia
Brief Title: Home Away From Home - Medical Outcomes
Acronym: Aim 1
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: C.S. Mott Children's Hospital (Other); Children's Healthcare of Atlanta (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Medical Center Dallas (Other); Children's Hospital of Michigan (Other); Baylor College of Medicine (Other); University of Mississippi Medical Center (Other); Arkansas Children's Hospital Research Institute (Other); Ochsner Health System (Other); Lucile Packard Children's Hospital (Other); Primary Children's Hospital (Other); Rady Children's Hospital, San Diego (Other); Seattle Children's Hospital (Other); Patient-Centered Outcomes Research Institute (Other); Children's Hospital Colorado (Other); Alfred I. duPont Hospital for Children (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-012074
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Acute Myeloid Leukemia; Neutropenia; Bacteremia
Keywords: Pediatric; Neutropenia Management; Acute Myeloid Leukemia; Chart Abstraction; Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neutropenia; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Discharge Management: Discharge to outpatient management during neutropenia within 3 days after chemotherapy completion in a given course
- Inpatient Management: Remain hospitalized during chemotherapy-induced neutropenia

SUMMARY:
Treatment for pediatric acute myeloid leukemia (AML) involves intensive chemotherapy regimens that result in periods of profound neutropenia leaving patients susceptible to severe infectious complications. Infectious complications are the leading cause of treatment related mortality among AML patients, but there are little clinical data to inform whether management of neutropenia post AML chemotherapy should occur in an outpatient or inpatient setting. The primary objective of this study is to compare the clinical effectiveness of outpatient versus inpatient management of neutropenia in children with AML.

DETAILED DESCRIPTION:
This is a bidirectional observational cohort study.

Participants will be patients less that 19 years of age at diagnosis receiving or having received chemotherapy for AML from seventeen participating pediatric hospitals across the United States. There is no study intervention; this is a medical record abstraction study only. Investigators will abstract subjects medical record data over the study period in order to study clinical outcomes including the occurrence of bacteremia and time to the start of the next course in the chemotherapy regimen, in relation to neutropenia management strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of age less than 19 at diagnosis.
2. Receipt or planned receipt of AML chemotherapy between January 1, 2012 and December 31, 2019.

Exclusion Criteria:

1. Patients being treated for relapsed AML
2. Patients with Acute Promyelocytic Leukemia (APML)
3. Patients undergoing stem cell transplant (SCT)
4. Patients receiving reduced intensity frontline chemotherapy

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include all AML patients who received or will receive chemotherapy between January 1, 2012 and December 31, 2019 at any of the fifteen participating pediatric institutions across the US. Patients discharged within 3 days after completion of that chemotherapy course will be categorized as 'early discharge' to outpatient management during neutropenia. Patients meeting eligibility criteria for 'early discharge' but remaining in the hospital more than 3 days after completion of that chemotherapy course will be categorized as inpatient management. Patients will be considered early discharge-eligible if there is no evidence of fever, infection or intensive care unit (ICU) level care within ± 3 days of the last dose of chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2015-06; Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (17):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Dana-Farber Cancer Institute/Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Coded, limited data sets will be shared with participating sites upon approved request. Only aggregate level data will be shared with the study sponsor Patient-Centered Outcomes Research Institute (PCORI).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 610 patients reflects the total number of patients included in chart abstractions; from there exclusion criteria were applied to determine early discharge eligibility. They were assigned to Early Discharge Management and Inpatient Management by chemotherapy course, not by the overall treatment.
Groups:
- Pediatric AML Patients: All patients included in chart abstractions. Exclusion criteria were applied to these patients to determine if they were early discharge eligible. Then they were assigned to outpatient-managed and inpatient-managed arms.
Period: Overall Study
Arm/Group | Pediatric AML Patients
Started | 610
Induction I (Patients whose Induction I course was included in chart abstractions.) | 585
Early Discharge Eligible at Induction I (Study population after early discharge criteria were applied at Induction I.) | 276 (24 of these patients were managed as outpatients. 252 were managed as inpatients.)
Induction II (Patients whose Induction II course was included in chart abstractions.) | 564
Early Discharge Eligible at Induction II (Study population after early discharge criteria were applied at Induction II.) | 493 (114 of these patients were managed as outpatients. 379 were managed as inpatients.)
Intensification I (Patients whose Intensification I course was included in chart abstractions.) | 476
Early Discharge Eligible at Int I (Study population after early discharge criteria were applied at Intensification I.) | 374 (104 of these patients were managed as outpatients. 270 were managed as inpatients.)
Intensification II (Patients whose Intensification II course was included in chart abstractions.) | 342
Early Discharge Eligible at Int II (Study population after early discharge criteria were applied at Intensification II.) | 285 (56 of these patients were managed as outpatients. 229 were managed as inpatients.)
Intensification III (Patients whose Intensification III course was included in chart abstractions.) | 48
Early Discharge Eligible at Int III (Study population after early discharge criteria were applied at Intensification III.) | 44 (7 of these patients were managed as outpatients. 37 were managed as inpatients.)
Completed (This milestone reflects the total early discharge-eligible study population in the overall study.) | 575
Not Completed | 35

BASELINE CHARACTERISTICS:
Population: These were the discharge eligible patients who either remained inpatient or were managed outpatient during study course Induction II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Discharge Management | Inpatient Management | Total
Number analyzed (Participants) | 114 | 379 | 493
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 114 | 379 | 493
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 192 | 245
  Male | 61 | 187 | 248
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 52 | 224 | 276
  Race: Black | 17 | 74 | 91
  Race: Asian | 11 | 26 | 37
  Race: Other | 33 | 44 | 77
  Race: Not recorded in EMR | 1 | 11 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity: Hispanic Ethnicity | 29 | 77 | 106
  Hispanic Ethnicity: Not Hispanic Ethnicity | 85 | 302 | 387
Region of Enrollment [Number; unit: participants]
  United States | 114 | 379 | 493

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Post-chemotherapy Bacteremia
Description: Identification of bacteremia will begin three days after completion of a chemotherapy course and will continue until recovery of absolute neutrophil count (ANC > 200 uL), or until the start of the next course (for a very small number of patients who begin the next course of chemotherapy prior to count recovery). Bacteremia will be defined as a single positive blood culture for a bacterial pathogen (including Viridans group Streptococci). If the bacterium is an organism considered as a common commensal organism by the National Healthcare Safety Network, two separate positive blood cultures will be required for classification as bacteremia.
Time Frame: Identification of bacteremia will begin three days after completion of a chemotherapy course and will continue until recovery of absolute neutrophil count (ANC > 200 uL), or until the start of the next course.
Population: Patients in study course Induction II analyzed for bacteremia for this course.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Discharge Management | Inpatient Management
Number analyzed (Participants) | 114 | 379
Participants | 22 | 81

2. Secondary Outcome: Time to the Initiation of the Next Chemotherapy Course
Description: Time to next course of chemotherapy will be measured as the number of days from the three days after the completion chemotherapy in a given course until the first day of the next course.
Time Frame: The number of days from the three days after the completion chemotherapy in a given course until the first day of the next course
Population: Patients in Induction II who were analyzed for the amount of time (in days) it took for them to start their next chemotherapy course.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Discharge Management | Inpatient Management
Number analyzed (Participants) | 114 | 379
days | 31.5 (9.4) | 27.8 (7.6)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored while chart abstractions began in December 2015 and were completed in July 2019. As this is an observational study, it was determined that adverse events were a non-issue.
Description: There is no study intervention; this is a medical record abstraction study only, thus adverse events were not monitored or assessed.
Arm/Group | Early Discharge Management | Inpatient Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02774850/Prot_SAP_000.pdf